CLINICAL TRIAL: NCT02814435
Title: Quality of Life Measures in Patients With Retinal Degeneration
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: QoLMeasuresIRD
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Retinal Degeneration
Keywords: Retina; Retinal Degeneration; Quality of Life Measures
MeSH Terms: conditions — Retinal Degeneration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with inherited retinal degeneration will answer two questionnaires and undergo a computerised contrast sensitivity function test.
  Interventions: Other: Questionnaire; Other: Computerised contrast sensitivity function test
- Normal controls: Normal controls recruited by advertising will answer two questionnaires and undergo a computerised test that assess contrast sensitivity function.
  Interventions: Other: Questionnaire; Other: Computerised contrast sensitivity function test

INTERVENTIONS:
Other: Questionnaire — The participants will answer two questionnaires. These are the NEI VFQ-25 and the DLTV (daily living tasks of vision).
Other: Computerised contrast sensitivity function test — This test involves the patient identifying whether bars on a screen are horizontal or vertical. It is designed to measure contrast sensitivity.

SUMMARY:
Inherited retinal degeneration (IRD) is a major cause of blindness and partial loss of vision cases in the UK and starts at an early age. The purpose of this observational study is to use the results of two questionnaires and a computerised test testing contrast sensitivity, to assess the impact of IRD on quality of life. This study will involve collecting data from patients with IRD, but also collecting data from normal controls.

DETAILED DESCRIPTION:
IRD presents a significant burden on the NHS as well as on the individual and families. IRDs are particularly difficult in a family situation due to guilt and other complex emotions related to inheritance patterns. Poorer mental health has been reported in patients with retinitis pigmentosa, manifesting in a range of ways including stress, depression and anxiety, particularly as the disease progresses. This is most probably caused by the uncertainty of the disease process and the progressive nature of the degeneration.

Recent work has reported that quality of life significantly deteriorates with a drop in visual field diameter of 20 degrees or a drop in visual acuity lower then LogMAR 0.3 (equivalent to 6/12). Contrast sensitivity is often used in conjunction with VA to assess visual capabilities. It is a measure of the ability to see reduced contrast and has a major impact on utility of vision. Relating contrast sensitivity function to quality of life will provide valuable information about whether this aspect of vision is a critical measure for patient health. This is especially important as novel treatments are being developed for the treatment of IRDs.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing & able to give informed consent for participation in the study.
* Male or female, aged 18 - 85.
* A clinical or genetic diagnosis of retinal degeneration or normal age and sex-matched controls without known retinal disease.
* Able to participate in visual function testing.

Exclusion Criteria:

* The participant may not enter the study if any of the following apply:

  * 1) they have a pre-existing amblyopia or squint;
  * 2) they have any other retinal problems that may confound the measures assessed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with inherited retinal degeneration will be recruited from the outpatient clinic in the Oxford Eye Hospital. 30 healthy controls will be recruited from advertising around the OUH hospitals and the University of Oxford.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Impact of inherited retinal degeneration on quality of life measures. | May 2016 to May 2017
  This will be assessed by comparing questionnaire results between different inherited retinal degeneration types.This will be determined by using ANOVA testing to compare scores caused by different genetic mutations, allowing us to relate mutations causing central versus peripheral visual loss to the quality of life measures.

SECONDARY OUTCOMES:
Effect of contrast sensitivity function on quality of life. | May 2016 to May 2017
  Contrast sensitivity function will be related to the questionnaire results using ANOVA testing & correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jasleen K Jolly, MSc, Principal Investigator — University of Oxford
Locations (1):
- Oxford Eye Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ndcn.ox.ac.uk/divisions/nlo/